CLINICAL TRIAL: NCT03039855
Title: Tiara™ Transcatheter Mitral Valve Replacement Study (TIARA-II)
Brief Title: Tiara™ Transcatheter Mitral Valve Replacement Study
Acronym: TIARA-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 047-CPT-003
Record Dates: First submitted 2017-01-16; First posted 2017-02-01 (Estimated); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Mitral Valve Regurgitation
Keywords: Mitral; Regurgitation; Heart valve; Transcatheter; Transapical; Functional; Degenerative; TMVR
MeSH Terms: conditions — Mitral Valve Insufficiency; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Transcatheter mitral valve replacement with the TIARA valve and transapical delivery system
  Interventions: Device: TIARA valve and transapical delivery system

INTERVENTIONS:
Device: TIARA valve and transapical delivery system — Transcatheter mitral valve replacement
  Other Names: TIARA Mitral Transcatheter Heart Valve, TIARA Transapical Delivery System

SUMMARY:
To evaluate the safety and performance of the Neovasc Tiara Mitral Transcatheter Heart Valve with the Tiara Transapical Delivery System.

DETAILED DESCRIPTION:
The TIARA-II study is an international, multicenter, single-arm, prospective, safety and performance clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Severe mitral regurgitation
* High surgical risk for open mitral valve surgery
* Subject meets anatomical eligibility criteria

Exclusion Criteria:

* Deemed too frail by objective frailty assessments
* Previous cardiac procedures: any mitral valve replacement surgery and cardiac transplant
* Unsuitable cardiac structure
* Clinically significant untreated Coronary Artery Disease (CAD)
* Subjects on chronic dialysis
* Pregnant or planning pregnancy within next 12 months
* Documented bleeding or coagulation disorders
* Active infections requiring antibiotic therapy
* Subjects with a life expectancy less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Freedom from all-cause mortality | 30 days
Freedom from major adverse events | 30 Days
Reduction of Mitral Regurgitation to optimal or acceptable | 30 days

SECONDARY OUTCOMES:
Freedom from all-cause mortality | 90 days, 180 days, one year and annually to five years
Freedom from major adverse events | 90 days, 180 days, one year and annually to five years
Technical success | Day 0
  Per MVARC criteria
Procedural success | 30 days
  Per MVARC criteria
Device success | Day 0, Day 10, 30 days, 90 days, 180 days, one year and annually for five years
  Per MVARC criteria
NYHA Functional Class | 30 days, 90 days, 180 days and once annually for five years
  Number of subjects with improved NYHA class
6 Minute Walk Test | 30 days, 90 days, 180 days and once annually for five years
  Increase in distance (m) from baseline
Kansas City Cardiomyopathy Questionnaire | 30 days, 90 days, 180 days and once annually for five years
  Improvement in quality of life
Hemodynamic performance | 30 days, 90 days, 180 days and once annually for five years
  Assessed by echocardiography
Patient success | 1 year
  Per MVARC Criteria

CONTACTS AND LOCATIONS:
Locations (20):
- Germany (11):
  - Kerckhoff Klinik Herzzentrum-Herzchirurgie, Bad Nauheim
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Schüchtermann-Klinik, Bad Rothenfelde
  - Deutches Herzzentrum Berlin, Berlin
  - Immanuel Klinikum Bernau und Herzzentrum Brandenburg, Bernau
  - St.-Johannes-Hospital, Klinik für Innere Medizin I, Dortmund
  - Universitätsklinikum Halle, Halle
  - Universitasklinikum Hamburg-Eppendorf, Hamburg
  - Herzzentrum Leipzig, Leipzig
  - Herz-Kreislauf-Zentrum Klinikum Hersfeld Rotenburg, Rotenburg an der Fulda
  - Sana Herzchirurgie Stuttgart GmbH, Stuttgart
- Tel Aviv Medical Center, Tel Aviv, Israel
- Italy (4):
  - Fondazione Policlinico Universitario A. Gemelli - Università Cattolica del Sacro Cuore., Roma, RM
  - Fondazione Toscana 'Gabriele Monasterio', Massa
  - Ospedale San Raffaele, Milan
  - IRCCS Policlinico San Donato, San Donato Milanese
- St. Antonius Hospital, Nieuwegein, Netherlands
- Hospital Clinico San Carlos, Madrid, Spain
- United Kingdom (2):
  - Edinburgh Heart Centre Royal Infirmary, Edinburgh
  - King's College Hospital, London

REFERENCES:
- See also: Company website with product information — http://www.neovasc.com